CLINICAL TRIAL: NCT05734170
Title: The Effect of Chia Seeds on HDL Cholesterol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edward Via Virginia College of Osteopathic Medicine (Other)
Responsible Party: Principal Investigator, Brian Dickens, Principal Investigator, Discipline Chair for Family Medicine, Edward Via Virginia College of Osteopathic Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2015-011
Record Dates: First submitted 2022-11-21; First posted 2023-02-17 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Diet; Habits
Keywords: HDL; Cholesterol; Chia; Oats
MeSH Terms: conditions — Habits

STUDY DESIGN:
Intervention Model Description: This pilot study was a small, randomized controlled trial at an academic primary care center. Each patient provided voluntary written consent prior to participating in the project. At the beginning of the study, each participant was randomly assigned to the red, white or blue group. They were then assigned a number within that group. The red group was instructed to consume one serving of Cheerios according to package instructions each morning for 30 days, the white group one packet of instant oatmeal, and the blue group one packet of instant oatmeal with two tablespoons of chia seeds. Subjects will be questioned to ensure to contraindications to participation. All other dietary or exercise habits will be maintained to reduce risk of confounding variables.Cholesterol profiles and weight will be measured at the beginning and end of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cheerio breakfast (Other): Patient consumes 1 serving of cheerios for breakfast every day for 1 month. Blood is drawn to assess lipid panels before diet and after 1 month of diet.
  Interventions: Dietary Supplement: Cheerio Breakfast
- Instant Oatmeal Breakfast (Other): Patient consumes 1 package instant oatmeal for breakfast each day for 1 month. Blood is drawn to assess lipid panels before diet and after 1 month of diet.
  Interventions: Dietary Supplement: Instant Oatmeal breakfast
- Chia Seeds and Instant Oatmeal breakfast. (Experimental): Patient consumes 1 package instant oatmeal with 2 tbsp chia seeds everyday for breakfast for 1 month. Blood is drawn to assess lipid panels before diet and after 1 month of diet.
  Interventions: Dietary Supplement: Chia Seeds and instant oatmeal breakfast

INTERVENTIONS:
Dietary Supplement: Chia Seeds and instant oatmeal breakfast — The final group was to consume one packet of instant oatmeal with two tablespoons of chia seeds mixed in with oatmeal for breakfast for 30 days.
  Arms: Chia Seeds and Instant Oatmeal breakfast.
Dietary Supplement: Cheerio Breakfast — Patients were instructed to consume one serving of Cheerios according to package instructions each morning for 30 days.
  Arms: Cheerio breakfast
Dietary Supplement: Instant Oatmeal breakfast — The second group was assigned to consume one packet of instant oatmeal for 30 days.
  Arms: Instant Oatmeal Breakfast

SUMMARY:
The purpose of this clinical trial is to demonstrate the effect of daily consumption of chia seeds, if any, on HDL cholesterol levels and compare this to the effects of oats on HDL levels in adult populations.

DETAILED DESCRIPTION:
Chia seeds are touted as a health food capable of a beneficial effect on HDL cholesterol. Similar claims have been made for oats in various forms, claiming they improve cholesterol or are in some way heart healthy.

The investigators wish to demonstrate the effect of daily consumption of chia seeds, if any, on HDL cholesterol levels and compare this to the effects of oats on HDL levels.

This pilot study was a randomized controlled trial at an academic primary care center. Participation was voluntary and all participants provided written consent prior to enrollment. There were no exclusionary criteria other than that participants must be adults willing to come in to get their cholesterol profiles checked at the beginning and end of the study. Participants consumed their assigned breakfast in a standard serving size for a month with blood draws and weights recorded before and after the diet. Patients' cholesterol profiles were also compared with their weights. To standardize the delivery of chia seeds, the group consuming chia seeds mixed the chia with oatmeal. The three groups thus consisted of Cheerios, oatmeal and oatmeal with chia seeds. Initially, there were a total of 11 subjects, three in the Cheerios group, four in the oatmeal group, and four in the oatmeal with chia seeds group. Two subjects were lost to follow-up, one each from the Cheerios and oatmeal groups, respectively. Statistical analysis including one way analysis was done with means, Wilcoxon/Kruskal Wallis test and 1 way test.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to give voluntary consent
* Must be greater than or equal to 18 years old
* Must be willing to give blood twice
* Must be able to eat assigned breakfast

Exclusion Criteria:

* "Subjects between the ages of 18 and 50 years old without a history of food allergies to either chia seeds or oats, kidney stones or a history of hyperlipidemia or treatment for hyperlipidemia will be eligible."

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-07-28 (Actual); Primary Completion 2015-08-27 (Actual); Study Completion 2015-08-27 (Actual)

PRIMARY OUTCOMES:
Lipid Panel | 1 month
  Patients' blood was taken twice with intent to measure the cholesterol profile, including: total triglycerides, LDL cholesterol, and HDL cholesterol.

SECONDARY OUTCOMES:
Weight | 1 month
  Patients' weight will be taken twice. Once before the diet and once upon completion of the diet.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: The promising future of chia, Salvia hispanica L — http://pubmed.ncbi.nlm.nih.gov/23251075/
- See also: Dietary levels of chia: influence on yolk cholesterol, lipid content and fatty acid composition for two strains of hens — https://pubmed.ncbi.nlm.nih.gov/10824962/
- See also: EFFECT OF CHIA SEED (SALVIA HISPANICA L.) CONSUMPTION ON CARDIOVASCULAR RISK FACTORS IN HUMANS: A SYSTEMATIC REVIEW — https://pubmed.ncbi.nlm.nih.gov/26545644/
- See also: Diet-induced oxalate nephropathy from excessive nut and seed consumption — https://casereports.bmj.com/content/13/11/e237212
- See also: A dietary pattern including nopal, chia seed, soy protein, and oat reduces serum triglycerides and glucose intolerance in patients with metabolic syndrome — https://pubmed.ncbi.nlm.nih.gov/22090467/